CLINICAL TRIAL: NCT02263170
Title: Assessment of Anatomic, Physiologic and Biomechanical Characteristics of the Anal Canal and Pelvic Floor. An Observational Pilot Study
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Nano-Tera.ch, Lausanne (Unknown); Spitäler Schaffhausen (Unknown); University of Bern (Other); University of Basel (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-BE: 048/2014
Record Dates: First submitted 2014-10-01; First posted 2014-10-13 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence | interventions — Magnetic Resonance Spectroscopy; CASP8 and FADD-Like Apoptosis Regulating Protein

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- All study participants: Healthy (m/f), normal weighted
  Interventions: Other: MRI (magnetic resonance imaging); Other: US (ultra sound); Other: FLIP (functional luminal imaging probe); Other: HRAM (high resolution anal manometry)

INTERVENTIONS:
Other: MRI (magnetic resonance imaging) — Assessment of the sphincter morphology
Other: US (ultra sound) — Assessment of the sphincter morphology
Other: FLIP (functional luminal imaging probe) — Assessment of the biomechanical properties of the sphincter region
Other: HRAM (high resolution anal manometry) — Assessment of the biomechanical properties of the sphincter region

SUMMARY:
With the project Smart Muscle for Incontinence Treatment (SMIT) a multidisciplinary consortium consisting of representatives ranging from clinical medicine via microelectronics towards biomaterial science aims to develop a novel implant to treat faecal incontinence. The aim of this campaign includes development of implantable prototype devices acting as artificial continence muscles using low-voltage electrically activated polymers (EAPs) controlled by implemented pressure sensors and the patient.

Subsequently, the knowledge of the anatomical and biomechanical properties of the anal sphincter complex are of cardinal importance. Most of the existing data on anatomy and physiology results is based on old studies and almost no data on biomechanical properties are available. However, new technologies or even merging data from different examination methods might provide new information in this field.

DETAILED DESCRIPTION:
Background

Fecal incontinence (FI) is affecting self-confidence and can lead to social isolation and even loss of employment Often conservative treatment as the first option is ineffective and surgical interventions follow conservative are necessary.

Small defects of the anal sphincter muscles might be treated with sphincter repair and sacral neuromodulation (SNM) However, patients rarely become fully continent or short-term results deteriorate in the long term [1]. Those patients and patients with large defects are candidates for a neosphincter procedure (artificial bowel sphincter or graciloplasty). However, the success rate of these methods is limited and the explantation rate is high. A permanent colostomy associated with massive psychosocial impairment remains as ultimate treatment option With the project Smart Muscle for Incontinence Treatment (SMIT) a multidisciplinary consortium consisting of representatives ranging from clinical medicine via microelectronics towards biomaterial science aims to develop a novel implant to treat faecal incontinence. The aim of this campaign includes development of implantable prototype devices acting as artificial continence muscles using low-voltage electrically activated polymers (EAPs) controlled by implemented pressure sensors and the patient.

Subsequently, the knowledge of the anatomical and biomechanical properties of the anal sphincter complex are of cardinal importance. Most of the existing data on anatomy and physiology results is based on old studies and almost no data on biomechanical properties are available. However, new technologies or even merging data from different examination methods might provide new information in this field.

Accurate imaging data on the pelvic floor region is crucial for the development of a new, implantable device for restoration of fecal continence. Optimal size (inner, outer diameter, length) and geometrical shape (cylinder, cone, torus) adapted to different functional states (rest, squeezing, defecation) will improve function and prevent erosion and consequent infection of such a prosthesis.

With this study, the investigators aim to correlate three-dimensional endoanal ultrasonographic images with MRI images. The combination of different imaging techniques has been demonstrated to eliminate individual drawbacks of the examination methods and therefore would allow a precise description of the tissue [2]. The registered data with their complementary information would permit the distinct segmentation and three-dimensional presentations of the anatomical structures in the pelvic area. This information has a great potential to facilitate diagnostics and surgical planning in this region.

High-resolution anal manometry (HRAM) provides intra-anal pressure during rest or maximum pressure with high spatial and time resolution.

However Biomechanical properties of the anal canal as elasticity or stiffness (compliance or flexibility) of the tissue representing important parameters for a continence organ are not routinely evaluated in daily clinical practice. Functional Lumen Imaging Probe (FLIP) allows the measurement of a cross sectional area (CSA) with respect to applied luminal pressure, respectively. FLIP has the potential to be useful in order to assess the biomechanical properties of the sphincter region. Such information potentially gives new insights in physiology and pathophysiology of the continence process.

With this pilot study, the investigators aim to acquire anatomical and biomechanical data using established (manometry) and novel technologies (merging endoanal ultrasound and MRI data) in 20 healthy probands (10 male, 10 female).

Objective

Primary objective is to collect anatomical, physiological and biomechanical characteristics of the continence organ (sphincters and pelvic floor) in order to specify properties of a new implant for the treatment of faecal incontinence.

Secondary objectives are: test feasibility of FLIP in measuring the biomechanical properties of the anal canal and test feasibility of merging 3D US data and MR images.

Further this preliminary data will be used to plan an observational study comparing healthy probands and patients with incontinence.

Methods

For the assessment of the morphology ultra sound and MRI will be used, whereas FLIP (functional luminance imaging probe) and HRAM (high resolution anal manometry) are the modality of choice to investigate the biomechanical properties of the sphincter complex.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Absence of ano-rectal or pelvic floor symptoms (patient history, Wexner score and Longo's obstructed defecation syndrome (ODS) score =0. Appendix Constipation and Faecal Incontinence Score form)
* MRI safety (no metallic implants. Appendix MRI safety form)
* Normal weighted (20<BMI<30)
* Age ≥ 60 years

Exclusion Criteria

* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.)
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* age (<18 years old)
* history of complicated child delivery
* previous anorectal surgery

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited by flyers and advertisement in internet.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Sphincter morphology | At baseline
  Functional sphincter variables are: anal canal length, resting, squeeze, and relaxation pressures, squeeze time, anal pressure in response to coughing, RAIR (percentage of anal relaxation), rectal volume filling to first sensation, urge and maximal tolerable volume, and distension of the anal canal in response to different filling volumes. Anatomical parameters are: distinction between internal and external sphincter (yes/no), sphincter lengths, sphincter thickness, and sphincter volumes.

SECONDARY OUTCOMES:
Test feasibility of FLIP in measuring the biomechanical properties of the anal canal | At baseline
  Test the ability of FLIP in order to assess the biomechanical properties of the human anal sphincter complex in sufficient quality
Test feasibility of merging 3D US data and MR images | At baseline
  Test feasibility of merging 3D US data and 3D MR images (full body MR and endoanal coil MR) in order to get a more precise anatomical image at once

CONTACTS AND LOCATIONS:
Overall Officials: Bert Müller, Prof. Dr., Study Director — Biomaterials Science Center (BMC) University of Basel c/o University Hospital Basel 4031 Basel
Locations (1):
- Universitätsklinik für Viszerale Chirurgie und Medizin Bauchzentrum Bern (Inselspital Bern), Bern, Switzerland

REFERENCES:
- See also: Related Info — http://www.nano-tera.ch/projects/341.php